CLINICAL TRIAL: NCT06865443
Title: Evaluation of CD47, "Do Not Eat Me" Signal Expression in Chronic Myeloid Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Ehab Fawzy Abdou, residant doctor, Assiut University
Other Study IDs: CD47 Chronic Myeloid Leukemia
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: CML patients, who fulfill the WHO 2022 criteria

SUMMARY:
Chronic myeloid leukemia is a myeloid neoplasm characterized by the overproduction of mature granulocytes . Cluster of differentiation 47 (CD47) is a membrane protein, which is over-expressed by virtually all cancers and regulates many signaling systems associated with tumor growth and invasion. Following CD47 binding to the inhibitory receptor (signal regulatory protein, SIRPα) on macrophages, the CD47-receptor complex sends a "do not eat me" anti-phagocytic signal to prevent phagocytosis . This balance is tipped by cancer cells, which adopt the "self" signal and upregulate CD47 expression to evade immune surveillance and subsequent destruction. Elevated expression of CD47 has been observed in ovarian carcinoma cell lines , murine myeloid leukemias , leukemic stem cells and several solid tumors .

Flow cytometry revealed high surface expression of CD47 on 73% of samples collected from the bone marrow of multiple myeloma (MM) patients .

High CD47 expression on six different primary effusion lymphoma (PEL) cell lines compared to peripheral blood mononuclear cells (PBMC) was found . Additionally, in acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), and several non-Hodgkin's lymphoma (NHL) subtypes, increased CD47 expression is correlated with adverse clinical outcomes .

Hematological malignancies, even at onset, present with widespread bone marrow and peripheral blood involvement and many are still without effective systemic curative therapies . Most CML patients have deep and durable responses when treated with BCR::ABL1 tyrosine kinase inhibitors, which might be influenced by long-term toxicities during the treatment .

CD47 "don't eat me signal" expression not evaluated in CML. the aim of the study To detect CD47 expression by flow cytometry in CML patients. To study the correlation between BCR::ABL1 gene and CD47 expression in CML patients . Evaluation of the role CD47 as predictor of CML patient outcome

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* both sex
* CML patients, who fulfill the WHO 2022 criteria

Exclusion Criteria:

* Patients with other haematological neoplasms (ALL,CLL, plasma cell myeloma)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: CML patients, who fulfill the WHO 2022 criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
CD47 Signal Expression in Chronic Myeloid Leukemia | baseline
  CD47 Signal Expression in Chronic Myeloid Leukemia